CLINICAL TRIAL: NCT00036270
Title: Randomized Phase III Study Of Exemestane (Aromasin) For 5 Years Versus Tamoxifen For 2.5- 3 Years Followed By Exemestane (Aromasin) For A Total Of 5 Years As Adjuvant Therapy For Postmenopausal, Receptor Positive, Node Negative or Node Positive Breast Cancer Patients
Brief Title: Randomized Phase III Study Of Exemestane (Aromasin) For 5 Years Versus Tamoxifen for 2.5 to 3 Years Followed By Exemestane
Acronym: TEAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 971-ONC-0028-081; A5991026
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Results first posted 2009-12-04 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exemestane (Experimental)
  Interventions: Drug: exemestane (Aromasin)
- tamoxifen + exemestane (Experimental)
  Interventions: Drug: tamoxifen + exemestane

INTERVENTIONS:
Drug: exemestane (Aromasin) — exemestane, orally, 25 mg, for 5 years
  Other Names: aromasin
  Arms: exemestane
Drug: tamoxifen + exemestane — tamoxifen, 20 mg, orally, daily, 2-3 years; followed by exemestane, orally, 25 mg, for a total of 5 years of therapy
  Arms: tamoxifen + exemestane

SUMMARY:
To compare the effects of exemestane for 5 years versus tamoxifen and exemestane given sequentially over 5 years in the adjuvant treatment of postmenopausal women with early breast cancer.

This Pfizer sponsored trial is part of an international collaboration of investigators conducting 7 similar yet independent studies in 9 countries. This study is designed to be part of the larger TEAM trial where the data from these 7 studies will be combined. A pre-specified analysis of the pooled data will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed adenocarcinoma of the breast, followed by adequate surgical resection and/or radiotherapy, and/or adjuvant chemotherapy, if indicated.
* Stage T1-3 N0-2 Mo, Any TNM stage BC for whom adjuvant hormonal therapy is being considered.

Exclusion Criteria:

* Those patients not deemed to have had potentially curative primary surgical treatment or one of the following criteria:
* Inflammatory breast cancer
* Histologically positive supraclavicular nodes
* Ulceration/infiltration of local skin metastasis
* Neoadjuvant chemotherapy
* Ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) without invasion
* ER and PR negative primary tumor or ER/PR unknown status.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9779 (Actual)
Dates: Start 2001-08; Primary Completion 2008-10 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (142):
- United States (142):
  - Pfizer Investigational Site, Bessemer, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Flagstaff, Arizona
  - Pfizer Investigational Site, Green Valley, Arizona
  - Pfizer Investigational Site, Oro Valley, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Safford, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Sedona, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Tuscon, Arizona
  - Pfizer Investigational Site, North Little Rock, Arkansas
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Fort Collins, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Lone Tree, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Pueblo, Colorado
  - Pfizer Investigational Site, Thornton, Colorado
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Hudson, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Lauderhill, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orange Park, Florida
  - Pfizer Investigational Site, Palatka, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Saint Augustine, Florida
  - Pfizer Investigational Site, Alton, Illinois
  - Pfizer Investigational Site, Arlington Heights, Illinois
  - Pfizer Investigational Site, Niles, Illinois
  - Pfizer Investigational Site, Winfield, Illinois
  - Pfizer Investigational Site, Carmel, Indiana
  - Pfizer Investigational Site, Fishers, Indiana
  - Pfizer Investigational Site, Greenfield, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Shelbyville, Indiana
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Cedar Rapids, Iowa
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Shawnee Mission, Kansas
  - Pfizer Investigational Site, Westminster, Maryland
  - Pfizer Investigational Site, North Adams, Massachusetts
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Burnsville, Minnesota
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Maplewood, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Woodbury, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Lee's Summit, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Santa Fe, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Amsterdam, New York
  - Pfizer Investigational Site, Brockport, New York
  - Pfizer Investigational Site, Canandaigua, New York
  - Pfizer Investigational Site, Geneva, New York
  - Pfizer Investigational Site, Hudson, New York
  - Pfizer Investigational Site, Latham, New York
  - Pfizer Investigational Site, Rexford, New York
  - Pfizer Investigational Site, Troy, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Elizabeth City, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Kernersville, North Carolina
  - Pfizer Investigational Site, Lexington, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Seneca, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Bartlesville, Oklahoma
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Springfield, Oregon
  - Pfizer Investigational Site, Tualatin, Oregon
  - Pfizer Investigational Site, Kingston, Pennsylvania
  - Pfizer Investigational Site, Easley, South Carolina
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Abilene, Texas
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Bedford, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Denton, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Fredericksburg, Texas
  - Pfizer Investigational Site, Garland, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Kerrville, Texas
  - Pfizer Investigational Site, Lewisville, Texas
  - Pfizer Investigational Site, Longview, Texas
  - Pfizer Investigational Site, McAllen, Texas
  - Pfizer Investigational Site, Mesquite, Texas
  - Pfizer Investigational Site, Midland, Texas
  - Pfizer Investigational Site, New Braunfels, Texas
  - Pfizer Investigational Site, Odessa, Texas
  - Pfizer Investigational Site, Paris, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Round Rock, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Sherman, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Waco, Texas
  - Pfizer Investigational Site, Webster, Texas
  - Pfizer Investigational Site, Weslaco, Texas
  - Pfizer Investigational Site, Wichita Falls, Texas
  - Pfizer Investigational Site, Chesapeake, Virginia
  - Pfizer Investigational Site, Christianburg,, Virginia
  - Pfizer Investigational Site, Christianburg, Virginia
  - Pfizer Investigational Site, Fairfax, Virginia
  - Pfizer Investigational Site, Gainesville, Virginia
  - Pfizer Investigational Site, Hampton, Virginia
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Pulaski, Virginia
  - Pfizer Investigational Site, Roanoke, Virginia
  - Pfizer Investigational Site, Salem, Virginia
  - Pfizer Investigational Site, Williamsburg, Virginia
  - Pfizer Investigational Site, Woodbridge, Virginia
  - Pfizer Investigational Site, Wytheville, Virginia
  - Pfizer Investigational Site, Burien, Washington
  - Pfizer Investigational Site, Edmonds, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Vancouver, Washington

REFERENCES:
- [Derived] Leblanc A, Beltran-Bless AA, Pond GR, El Emam K, Juwara L, Clemons L, Bayani J, Pilgram L, Pharoah P, Mallon E, Taylor KJ, Markopoulos C, Dirix L, Vandermeer L, Hilton J, Savard MF, Bartlett JMS, Clemons M. Prognostic and predictive performance of PREDICT 2.1, PREDICT v3, and RSClin in node-negative early breast cancer: a TEAM pathology substudy. Breast Cancer Res Treat. 2026 Feb 5;215(3):74. doi: 10.1007/s10549-026-07909-5. PMID 41642493
- [Derived] Bayani J, Kornaga EN, Crozier C, Jang GH, Bathurst L, Kalatskaya I, Trinh QM, Yao CQ, Livingstone J, Boutros PC, Spears M, McPherson JD, Stein LD, Rea D, Bartlett JMS. Identification of Distinct Prognostic Groups: Implications for Patient Selection to Targeted Therapies Among Anti-Endocrine Therapy-Resistant Early Breast Cancers. JCO Precis Oncol. 2019 Dec;3:1-13. doi: 10.1200/PO.18.00373. PMID 35100692
- [Derived] Noordhoek I, Blok EJ, Meershoek-Klein Kranenbarg E, Putter H, Duijm-de Carpentier M, Rutgers EJT, Seynaeve C, Bartlett JMS, Vannetzel JM, Rea DW, Hasenburg A, Paridaens R, Markopoulos CJ, Hozumi Y, Portielje JEA, Kroep JR, van de Velde CJH, Liefers GJ. Overestimation of Late Distant Recurrences in High-Risk Patients With ER-Positive Breast Cancer: Validity and Accuracy of the CTS5 Risk Score in the TEAM and IDEAL Trials. J Clin Oncol. 2020 Oct 1;38(28):3273-3281. doi: 10.1200/JCO.19.02427. Epub 2020 Jul 24. PMID 32706636
- [Derived] Derks MGM, Bastiaannet E, van de Water W, de Glas NA, Seynaeve C, Putter H, Nortier JWR, Rea D, Hasenburg A, Markopoulos C, Dirix LY, Portielje JEA, van de Velde CJH, Liefers GJ. Impact of age on breast cancer mortality and competing causes of death at 10 years follow-up in the adjuvant TEAM trial. Eur J Cancer. 2018 Aug;99:1-8. doi: 10.1016/j.ejca.2018.04.009. Epub 2018 Jun 6. PMID 29885375
- [Derived] Bartlett JM, Brookes CL, Piper T, van de Velde CJ, Stocken D, Lyttle N, Hasenburg A, Quintayo MA, Kieback DG, Putter H, Markopoulos C, Kranenbarg EM, Mallon EA, Dirix LY, Seynaeve C, Rea DW. Do type 1 receptor tyrosine kinases inform treatment choice? A prospectively planned analysis of the TEAM trial. Br J Cancer. 2013 Oct 29;109(9):2453-61. doi: 10.1038/bjc.2013.609. Epub 2013 Oct 3. PMID 24091623
- [Derived] van de Velde CJ, Rea D, Seynaeve C, Putter H, Hasenburg A, Vannetzel JM, Paridaens R, Markopoulos C, Hozumi Y, Hille ET, Kieback DG, Asmar L, Smeets J, Nortier JW, Hadji P, Bartlett JM, Jones SE. Adjuvant tamoxifen and exemestane in early breast cancer (TEAM): a randomised phase 3 trial. Lancet. 2011 Jan 22;377(9762):321-31. doi: 10.1016/S0140-6736(10)62312-4. PMID 21247627
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=971-ONC-0028-081

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane: Exemestane (Aromasin®) 25 milligram (mg) once daily (QD) for 5 years.
- Tamoxifen Followed by Exemestane: Tamoxifen 20 mg QD; upon completing 2.5 years to 3 years of tamoxifen, participants were to be switched to exemestane 25 mg QD and then were to complete a total of 5 years endocrine therapy.
Period: Randomized to Study Treatment
Arm/Group | Exemestane | Tamoxifen Followed by Exemestane
Started | 4904 | 4875
Completed | 4898 | 4868
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 6 | 7
Period: Study Treatment to 5 Year Report
Arm/Group | Exemestane | Tamoxifen Followed by Exemestane
Started | 4898 | 4868
Treated | 4852 | 4814
Completed | 2333 | 1380
Not Completed | 2565 | 3488
Not completed — Ongoing | 1081 | 736
Not completed — Disease- Free Survival (DFS) event | 507 | 447
Not completed — Adverse Event | 501 | 782
Not completed — Other | 277 | 288
Not completed — Treatment refusal | 113 | 208
Not completed — Randomized but not treated | 46 | 54
Not completed — Protocol Violation | 23 | 91
Not completed — Intercurrent illness | 17 | 29
Not completed — Too early switch | 0 | 103
Not completed — No/too late switch/refusal to switch | 0 | 750

BASELINE CHARACTERISTICS:
Groups:
- Exemestane: Exemestane (Aromasin®) 25 mg QD for 5 years.
- Total: Total of all reporting groups
Arm/Group | Exemestane | Tamoxifen Followed by Exemestane | Total
Number analyzed (Participants) | 4898 | 4868 | 9766
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65 (9) | 64 (9) | 64 (9)
Age, Customized [Number; unit: Participants]
  Less than 50 years | 171 | 160 | 331
  50 to 59 years | 1510 | 1507 | 3017
  60 to 69 years | 1835 | 1896 | 3731
  Greater than and equal to 70 years | 1382 | 1305 | 2687
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4898 | 4868 | 9766
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS): Number of Events (Disease Relapse or Death) From Baseline up to 2.75 Years
Description: Number of events (disease relapse or death) to time of observation for DFS. DFS defined as time from randomization to earliest documentation of disease relapse or death from any cause in postmenopausal, receptor positive, node negative or node positive breast cancer patients for adjuvant treatment with exemestane compared with adjuvant tamoxifen therapy at 2.75 years. Disease relapse: primary tumor recurrence (locoregional or distant) and ipsilateral or contralateral breast cancer (CBC). Intercurrent death: death without disease relapse.
Time Frame: Baseline (Month 0) up to 2.75 years
Population: Intent-to-Treat (ITT) population: participants randomized to one of the two study arms (all randomized participants); (n) = number of participants at observation for exemestane and tamoxifen, respectively. All participants were censored at 2.75 years.
Measure: Number; unit: Events (disease relapse or death)
Arm/Group | Exemestane | Tamoxifen Followed by Exemestane
Number analyzed (Participants) | 4898 | 4868
Events (disease relapse or death) | 352 | 388
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen Followed by Exemestane; Analysis at 2.75 years post-randomization. Null hypothesis: no difference in DFS between the two treatments for the first 2.75 years. To maintain overall alpha of 0.05, 2 adjustments made: first, a nominal alpha of 0.0302 was used for the primary endpoint. Second, level of significant was 0.0012 for interim analysis; Test type: Superiority or Other; p = 0.118, Log Rank; Log rank (Mantel-Cox). Adjusted for overall stratification factor; 1 degree of freedom; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.77 to 1.03] — A hazard ratio less than 1 favors the test treatment (exemestane only arm)

2. Primary Outcome: Disease Free Survival (DFS): Number of Events (Disease Relapse or Death) From Baseline up to 5 Years
Description: Number of events (disease relapse or death) to time of observation for DFS. DFS defined as time from randomization to earliest documentation of disease relapse or death from any cause in postmenopausal, receptor positive, node negative or node positive breast cancer patients for adjuvant treatment with exemestane compared with adjuvant tamoxifen therapy at 5 years. Disease relapse: primary tumor recurrence (locoregional or distant) and ipsilateral or contralateral breast cancer (CBC). Intercurrent death: death without disease relapse.
Time Frame: Baseline (Month 0) up to 5 years
Population: ITT population included all participants who were randomized to one of the two study arms (all randomized participants); (n) = number of participants at observation for exemestane and tamoxifen, respectively. All participants were censored at the data cut off date of 08 November 2009.
Measure: Number; unit: Events (disease relapse or death)
Arm/Group | Exemestane | Tamoxifen Followed by Exemestane
Number analyzed (Participants) | 4898 | 4868
Events (disease relapse or death) | 712 | 714
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen Followed by Exemestane; Analysis at 5 years post-randomization. Null hypothesis: no difference in DFS between the two treatments for the first 5 years. To maintain overall alpha of 0.05, a nominal alpha of 0.0302 was used; Test type: Superiority or Other; p = 0.604, Log Rank; Log rank (Mantel-Cox). Adjusted for overall stratification factor; 1 degree of freedom; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.88 to 1.08] — A hazard ratio less than 1 favors the test treatment (exemestane only arm)

3. Secondary Outcome: Number of Events for Overall Survival (OS)
Description: Number of events (death) to time of observation for OS. OS is the duration from randomization to death. For participants who are alive, overall survival is censored at the last contact.
Time Frame: Baseline (Month 0) up to 5 years
Population: ITT population: participants randomized to one of the two study arms (all randomized participants); (n) = number of participants at observation for exemestane and tamoxifen, respectively. All participants were censored at the data cut off date of 08 November 2009.
Measure: Number; unit: Events (death)
Arm/Group | Exemestane | Tamoxifen Followed by Exemestane
Number analyzed (Participants) | 4898 | 4868
Events (death) | 485 | 476
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen Followed by Exemestane; Analysis at 5 years post-randomization. Null hypothesis: no difference in OS between the two treatments for the first 5 years. Overall alpha of 0.05 was maintained; Test type: Superiority or Other; p = 0.951, Log Rank; Log rank (Mantel-Cox). Adjusted for overall stratification factor; 1 degree of freedom; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.89 to 1.14] — A hazard ratio less than 1 favors the test treatment (exemestane only arm)

4. Secondary Outcome: Time to New Primary Breast Cancers
Description: New primary breast cancers were defined as events of ipsilateral/contralateral breast cancer (CBC).
Time Frame: Baseline (Month 0) up to 5 years
Population: Data was not analyzed due to insufficient number of events reported for the endpoint.
Arm/Group | Exemestane | Tamoxifen Followed by Exemestane
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Events for Time to Relapse
Description: Number of events to time of observation for relapse. Relapse is defined as all recurrences of the primary tumor (loco-regional and distant recurrence), second primary breast cancer, contralateral breast cancer.
Time Frame: Baseline (Month 0) up to 5 years
Population: as for outcome 3
Measure: Number; unit: Events (disease relapse)
Arm/Group | Exemestane | Tamoxifen Followed by Exemestane
Number analyzed (Participants) | 4898 | 4868
Events (disease relapse) | 499 | 521
Statistical Analysis 1: Comparison: Exemestane vs Tamoxifen Followed by Exemestane; Analysis at 5 years post-randomization. Null hypothesis: no difference in time to relapse between the two treatments for the first 5 years. Overall alpha of 0.05 was maintained; Test type: Superiority or Other; p = 0.293, Log Rank; Log rank (Mantel-Cox). Adjusted for overall stratification factor; 1 degree of freedom; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.83 to 1.06] — A hazard ratio less than 1 favors the test treatment (exemestane only arm)

6. Secondary Outcome: Number of Participants With New Primary Non-breast Cancers
Description: Number of participants with new primary non-breast cancers which included colorectal cancer, lung cancer, endometrial cancer, ductal carcinoma in situ (DCIS) and other primary cancer types.
Time Frame: Baseline (Month 0) up to 5 years
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Exemestane | Tamoxifen Followed by Exemestane
Number analyzed (Participants) | 4898 | 4868
Participants
  Colorectal cancer | 43 | 32
  Lung cancer | 24 | 17
  Endometrial cancer | 7 | 17
  DCIS | 3 | 4
  Other primary cancer types | 110 | 106

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tamoxifen Followed by Exemestane | Exemestane
Serious Adverse Events (participants affected / at risk) | 784/4814 | 831/4852
Other Adverse Events (participants affected / at risk) | 3551/4814 | 3567/4852
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen Followed by Exemestane (N=4814) | Exemestane (N=4852)
Anaemia (Blood and lymphatic system disorders) | 5 | 12
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 7 | 8
Angina unstable (Cardiac disorders) | 0 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 4
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 15 | 18
Atrial flutter (Cardiac disorders) | 1 | 2
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 4
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac asthma (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 7 | 9
Cardiac failure congestive (Cardiac disorders) | 6 | 12
Cardiac valve disease (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 2 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 2
Congestive cardiomyopathy (Cardiac disorders) | 1 | 1
Cor pulmonale (Cardiac disorders) | 1 | 2
Coronary artery disease (Cardiac disorders) | 7 | 8
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Cytotoxic cardiomyopathy (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 4
Mitral valve incompetence (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 18 | 18
Myocardial ischaemia (Cardiac disorders) | 1 | 4
Palpitations (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 5
Pleuropericarditis (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 2
Tachyarrhythmia (Cardiac disorders) | 0 | 3
Tachycardia (Cardiac disorders) | 4 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 | 1
Congenital musculoskeletal anomaly (Congenital, familial and genetic disorders) | 0 | 2
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1
Skull malformation (Congenital, familial and genetic disorders) | 1 | 0
Spine malformation (Congenital, familial and genetic disorders) | 3 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Otosclerosis (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 7 | 1
Goitre (Endocrine disorders) | 3 | 6
Hyperparathyroidism (Endocrine disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Thyroid disorder (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 1 | 1
Cataract (Eye disorders) | 2 | 3
Eye disorder (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 2 | 1
Retinal detachment (Eye disorders) | 0 | 3
Retinal disorder (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Retinal ischaemia (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Vitreous detachment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 11 | 14
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 1
Anal prolapse (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 3
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 10
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 4
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 6
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 4 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 6
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal tract irritation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 5 | 4
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mesenteric occlusion (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 5
Obstruction gastric (Gastrointestinal disorders) | 0 | 2
Oesophageal disorder (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 7 | 5
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Splenic artery aneurysm (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 6
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 3 | 6
Calcinosis (General disorders) | 1 | 0
Cardiac death (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 15 | 16
Condition aggravated (General disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Device breakage (General disorders) | 0 | 2
Device occlusion (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 4
Dysplasia (General disorders) | 0 | 1
Fat necrosis (General disorders) | 1 | 0
Fat tissue increased (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 4
Gait disturbance (General disorders) | 4 | 1
General physical health deterioration (General disorders) | 2 | 2
Hernia (General disorders) | 3 | 5
Hyperplasia (General disorders) | 3 | 1
Ill-defined disorder (General disorders) | 4 | 8
Impaired healing (General disorders) | 3 | 0
Implant site fibrosis (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Malaise (General disorders) | 3 | 1
Medical device complication (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Necrosis (General disorders) | 1 | 2
Nodule (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 1
Oedema due to cardiac disease (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 13 | 3
Polyp (General disorders) | 4 | 1
Pseudocyst (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 5
Sense of oppression (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 1
Swelling (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 13 | 11
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 10 | 14
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 4
Sarcoidosis (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 3 | 1
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 4 | 7
Appendicitis perforated (Infections and infestations) | 0 | 2
Arthritis bacterial (Infections and infestations) | 2 | 2
Bacterial infection (Infections and infestations) | 1 | 5
Breast abscess (Infections and infestations) | 4 | 2
Breast cellulitis (Infections and infestations) | 3 | 2
Breast infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 6 | 2
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 11 | 7
Cystitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 7 | 10
Endocarditis (Infections and infestations) | 0 | 1
Endometritis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 9 | 7
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 6 | 4
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 5 | 11
Lobar pneumonia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Lymphangitis (Infections and infestations) | 2 | 0
Mastitis (Infections and infestations) | 6 | 5
Meningitis (Infections and infestations) | 0 | 1
Molluscum contagiosum (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 26 | 25
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Post procedural cellulitis (Infections and infestations) | 2 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Pyoderma (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 10 | 4
Streptococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 6 | 7
Urosepsis (Infections and infestations) | 1 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 5 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 6 | 8
Breast injury (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 | 0
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 9
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 3
Femur fracture (Injury, poisoning and procedural complications) | 3 | 4
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 15 | 27
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 8
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 10
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 3 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 5
Poisoning (Injury, poisoning and procedural complications) | 1 | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation fibrosis (Injury, poisoning and procedural complications) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 4
Rib fracture (Injury, poisoning and procedural complications) | 2 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 2
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 3 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 4
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 5 | 6
Blood calcium increased (Investigations) | 0 | 1
Blood test abnormal (Investigations) | 0 | 1
CSF test abnormal (Investigations) | 1 | 0
Carbohydrate antigen 15-3 increased (Investigations) | 0 | 1
Clostridium test positive (Investigations) | 0 | 1
Coagulation test (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haemoglobin (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 0 | 1
Investigation (Investigations) | 0 | 1
Occult blood positive (Investigations) | 0 | 1
Prothrombin level increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 6
Enzyme abnormality (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 5
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 11 | 14
Arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 1
CREST syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 7
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 34
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Contralateral breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Dermatofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 8
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Mueller's mixed tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Paget's disease of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Alcoholic seizure (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 2 | 2
Apraxia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 3
Carotid artery thrombosis (Nervous system disorders) | 2 | 1
Carpal tunnel syndrome (Nervous system disorders) | 2 | 3
Cerebellar infarction (Nervous system disorders) | 0 | 2
Cerebral artery thrombosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 3 | 3
Cerebral infarction (Nervous system disorders) | 3 | 6
Cerebral ischaemia (Nervous system disorders) | 2 | 5
Cerebrovascular accident (Nervous system disorders) | 20 | 26
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 2
Coma (Nervous system disorders) | 1 | 3
Coma hepatic (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 2
Dementia (Nervous system disorders) | 0 | 2
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 5 | 4
Drop attacks (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 3
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 5
Hemiparesis (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
IIIrd nerve paresis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 2
Loss of consciousness (Nervous system disorders) | 1 | 3
Mental impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Myelitis transverse (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 1
Neuralgia (Nervous system disorders) | 1 | 3
Neuritis (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 2 | 2
Sedation (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 12 | 13
Thalamic infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 11 | 11
Alcohol abuse (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 4
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 10 | 9
Depression suicidal (Psychiatric disorders) | 2 | 0
Emotional distress (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 2
Calculus bladder (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Incontinence (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 4 | 7
Renal failure acute (Renal and urinary disorders) | 1 | 3
Renal infarct (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 4
Urinary retention (Renal and urinary disorders) | 1 | 1
Urogenital disorder (Renal and urinary disorders) | 2 | 0
Breast calcifications (Reproductive system and breast disorders) | 4 | 4
Breast cyst (Reproductive system and breast disorders) | 2 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 7
Breast enlargement (Reproductive system and breast disorders) | 1 | 2
Breast fibrosis (Reproductive system and breast disorders) | 1 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 1
Breast hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 3 | 4
Breast necrosis (Reproductive system and breast disorders) | 0 | 4
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 2
Cervical polyp (Reproductive system and breast disorders) | 4 | 0
Cystocele (Reproductive system and breast disorders) | 2 | 0
Endometrial atrophy (Reproductive system and breast disorders) | 2 | 0
Endometrial disorder (Reproductive system and breast disorders) | 2 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 17 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 3 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 3 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Nipple disorder (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 6 | 4
Ovarian disorder (Reproductive system and breast disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 3 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 3 | 1
Rectocele (Reproductive system and breast disorders) | 3 | 1
Urogenital prolapse (Reproductive system and breast disorders) | 1 | 0
Uterine atony (Reproductive system and breast disorders) | 1 | 0
Uterine disorder (Reproductive system and breast disorders) | 2 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 12 | 1
Uterine prolapse (Reproductive system and breast disorders) | 5 | 1
Vaginal disorder (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 9 | 4
Vaginal polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 3 | 1
Vulval disorder (Reproductive system and breast disorders) | 0 | 1
Vulval oedema (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal disorder (Reproductive system and breast disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 28
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22 | 24
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Scar (Skin and subcutaneous tissue disorders) | 1 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Alcohol detoxification (Surgical and medical procedures) | 0 | 1
Angioplasty (Surgical and medical procedures) | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 0 | 1
Arterial bypass operation (Surgical and medical procedures) | 1 | 0
Bile duct stent insertion (Surgical and medical procedures) | 1 | 0
Breast lump removal (Surgical and medical procedures) | 1 | 1
Breast operation (Surgical and medical procedures) | 2 | 2
Breast reconstruction (Surgical and medical procedures) | 3 | 2
Bunion operation (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1
Carpal tunnel decompression (Surgical and medical procedures) | 0 | 1
Cast application (Surgical and medical procedures) | 0 | 1
Cataract operation (Surgical and medical procedures) | 3 | 2
Cholecystectomy (Surgical and medical procedures) | 5 | 4
Cholelithotomy (Surgical and medical procedures) | 1 | 0
Colporrhaphy (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Drug therapy (Surgical and medical procedures) | 1 | 0
Eventration procedure (Surgical and medical procedures) | 1 | 0
Female genital operation (Surgical and medical procedures) | 1 | 2
Gastric bypass (Surgical and medical procedures) | 1 | 0
Gastric operation (Surgical and medical procedures) | 1 | 0
Haemangioma removal (Surgical and medical procedures) | 1 | 0
Hernia repair (Surgical and medical procedures) | 0 | 3
Hip arthroplasty (Surgical and medical procedures) | 4 | 10
Hip surgery (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 3 | 1
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Intervertebral disc operation (Surgical and medical procedures) | 0 | 1
Joint arthroplasty (Surgical and medical procedures) | 0 | 2
Knee arthroplasty (Surgical and medical procedures) | 7 | 4
Knee operation (Surgical and medical procedures) | 2 | 1
Lipoma excision (Surgical and medical procedures) | 0 | 1
Mastectomy (Surgical and medical procedures) | 4 | 1
Medical device removal (Surgical and medical procedures) | 1 | 0
Meniscus operation (Surgical and medical procedures) | 1 | 1
Meniscus removal (Surgical and medical procedures) | 0 | 1
Oophorectomy (Surgical and medical procedures) | 1 | 0
Osteosynthesis (Surgical and medical procedures) | 0 | 1
Phlebectomy (Surgical and medical procedures) | 0 | 1
Prolapse repair (Surgical and medical procedures) | 0 | 1
Radical hysterectomy (Surgical and medical procedures) | 1 | 0
Retinal operation (Surgical and medical procedures) | 1 | 0
Rotator cuff repair (Surgical and medical procedures) | 1 | 0
Scar excision (Surgical and medical procedures) | 1 | 1
Shoulder arthroplasty (Surgical and medical procedures) | 2 | 0
Simple mastectomy (Surgical and medical procedures) | 2 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 1
Spinal laminectomy (Surgical and medical procedures) | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 1
Tendon operation (Surgical and medical procedures) | 0 | 1
Thyroid nodule removal (Surgical and medical procedures) | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 0 | 5
Toe amputation (Surgical and medical procedures) | 1 | 0
Toe operation (Surgical and medical procedures) | 0 | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1 | 0
Uterine prolapse repair (Surgical and medical procedures) | 1 | 1
Vaginal operation (Surgical and medical procedures) | 0 | 1
Varicose vein operation (Surgical and medical procedures) | 0 | 2
Vascular operation (Surgical and medical procedures) | 0 | 1
Aneurysm (Vascular disorders) | 0 | 4
Aortic aneurysm (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 2 | 5
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 2
Arteritis (Vascular disorders) | 1 | 1
Circulatory collapse (Vascular disorders) | 1 | 3
Deep vein thrombosis (Vascular disorders) | 14 | 6
Embolism (Vascular disorders) | 4 | 2
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 3 | 0
Haemorrhage (Vascular disorders) | 2 | 1
Hot flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 6 | 11
Hypertensive crisis (Vascular disorders) | 0 | 8
Hypotension (Vascular disorders) | 0 | 2
Intermittent claudication (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 8 | 2
Shock (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 5 | 0
Thrombosis (Vascular disorders) | 13 | 6
Varicophlebitis (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 7
Vasculitis (Vascular disorders) | 1 | 0
Venoocclusive disease (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 6 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen Followed by Exemestane (N=4814) | Exemestane (N=4852)
Vertigo (Ear and labyrinth disorders) | 78 | 96
Abdominal pain (Gastrointestinal disorders) | 150 | 141
Constipation (Gastrointestinal disorders) | 274 | 236
Diarrhoea (Gastrointestinal disorders) | 258 | 302
Dry mouth (Gastrointestinal disorders) | 98 | 70
Dyspepsia (Gastrointestinal disorders) | 135 | 151
Nausea (Gastrointestinal disorders) | 482 | 419
Vomiting (Gastrointestinal disorders) | 106 | 96
Asthenia (General disorders) | 188 | 235
Chest pain (General disorders) | 91 | 100
Fatigue (General disorders) | 800 | 796
Oedema (General disorders) | 287 | 276
Oedema peripheral (General disorders) | 214 | 166
Pain (General disorders) | 492 | 541
Bronchitis (Infections and infestations) | 135 | 128
Cystitis (Infections and infestations) | 76 | 102
Herpes zoster (Infections and infestations) | 76 | 112
Infection (Infections and infestations) | 197 | 168
Nasopharyngitis (Infections and infestations) | 99 | 110
Urinary tract infection (Infections and infestations) | 114 | 129
Vaginal infection (Infections and infestations) | 100 | 47
Weight decreased (Investigations) | 140 | 187
Weight increased (Investigations) | 415 | 339
Decreased appetite (Metabolism and nutrition disorders) | 118 | 132
Hypercholesterolaemia (Metabolism and nutrition disorders) | 99 | 190
Hyperglycaemia (Metabolism and nutrition disorders) | 97 | 113
Arthralgia (Musculoskeletal and connective tissue disorders) | 1002 | 1157
Arthritis (Musculoskeletal and connective tissue disorders) | 130 | 161
Back pain (Musculoskeletal and connective tissue disorders) | 269 | 273
Bone pain (Musculoskeletal and connective tissue disorders) | 230 | 261
Muscle spasms (Musculoskeletal and connective tissue disorders) | 245 | 133
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 128 | 176
Myalgia (Musculoskeletal and connective tissue disorders) | 360 | 364
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 142 | 165
Osteoporosis (Musculoskeletal and connective tissue disorders) | 219 | 428
Pain in extremity (Musculoskeletal and connective tissue disorders) | 147 | 171
Amnesia (Nervous system disorders) | 143 | 188
Carpal tunnel syndrome (Nervous system disorders) | 76 | 109
Dizziness (Nervous system disorders) | 289 | 243
Headache (Nervous system disorders) | 372 | 369
Neuropathy peripheral (Nervous system disorders) | 120 | 174
Paraesthesia (Nervous system disorders) | 66 | 100
Anxiety (Psychiatric disorders) | 174 | 167
Depression (Psychiatric disorders) | 417 | 404
Insomnia (Psychiatric disorders) | 452 | 549
Libido decreased (Psychiatric disorders) | 164 | 196
Mood altered (Psychiatric disorders) | 147 | 151
Sleep disorder (Psychiatric disorders) | 61 | 110
Breast pain (Reproductive system and breast disorders) | 104 | 121
Vaginal discharge (Reproductive system and breast disorders) | 316 | 111
Vaginal haemorrhage (Reproductive system and breast disorders) | 186 | 94
Vulvovaginal dryness (Reproductive system and breast disorders) | 268 | 321
Cough (Respiratory, thoracic and mediastinal disorders) | 252 | 235
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 243 | 223
Alopecia (Skin and subcutaneous tissue disorders) | 299 | 329
Dry skin (Skin and subcutaneous tissue disorders) | 122 | 114
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 175 | 103
Night sweats (Skin and subcutaneous tissue disorders) | 102 | 87
Pruritus (Skin and subcutaneous tissue disorders) | 158 | 153
Rash (Skin and subcutaneous tissue disorders) | 216 | 227
Flushing (Vascular disorders) | 183 | 114
Hot flush (Vascular disorders) | 1690 | 1517
Hypertension (Vascular disorders) | 224 | 291
Lymphoedema (Vascular disorders) | 247 | 227

LIMITATIONS AND CAVEATS:
Overall Survival was reported as number of events which otherwise reported as time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.